CLINICAL TRIAL: NCT00059670
Title: Comparison of Two Therapies for UES Dysphagia
Brief Title: Comparison of Two Therapies for Upper Esophageal Sphincter (UES) Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: UESD (completed)
Record Dates: First submitted 2003-05-01; First posted 2003-05-02 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Deglutition Disorders
Keywords: UES; Dysphagia
MeSH Terms: conditions — Deglutition Disorders

INTERVENTIONS:
Procedure: Shaker Exercise vs. Traditional Dysphagia Therapy Regime

SUMMARY:
The aim of this research study is to determine the effectiveness of: 1) a traditional therapy regimen focusing on individual exercises for pharyngeal (throat) and laryngeal (voice box) musculature and 2) a new therapeutic exercise, the Shaker exercise.

The primary objective of this 5-year project is to identify which of two therapy programs, the Shaker exercise versus traditional therapy, results in the largest number of stable, non-oral dysphagic patients who can swallow safely and return to full oral feeding after 6 weeks of intervention. The study is powered adequately so that this aim can be tested separately for head and neck cancer and stroke patients. Our primary outcome measure is return to oral feeding, i.e., 100% of nutrition and hydration by mouth.

DETAILED DESCRIPTION:
Secondary aims of this research are:

1. Determine in a descriptive manner whether patients with residue in the pyriform sinuses who aspirate the residue after the swallow respond better, i.e., a higher percentage of them can return to 100% oral intake, than patients with residue in the valleculae who aspirate after the swallow or patients with residue in both locations who aspirate after the swallow and thus to define the spectrum of indications for the proposed exercise programs in the two groups of dysphagic patients (stroke and post-chemo radiation treatment for head and neck cancer) and whether postures enable each patient type to swallow more bolus types without aspiration at pre- and post
2. Define the pathophysiology underlying the swallow dysfunction and those pathophysiologic elements which change as a result of each therapy program including changes in -

   1. anteroposterior and lateral diameter of maximum deglutitive UES opening
   2. maximum deglutitive laryngeal anterior and superior excursions

ELIGIBILITY:
Inclusion Criteria (all required)

* Patients with pharyngeal phase dysphagia due to stroke or chemoradiation for head and neck cancer (without surgical intervention)
* Incomplete UES opening and post-deglutitive aspiration
* Hypopharyngeal (pyriform sinus) residue or vallecular residue alone or in combination
* Dysphagia requiring tube feeding (at least 3 months non-oral condition)
* Able to comply with protocol mandates, willing to perform the exercise programs, and ability to attend study sessions.

Exclusion Criteria

* Pharyngeal surgical procedures
* Other neuromuscular disorders such as
* Lack of cognition
* Metabolic myopathies
* History of alcoholic neuropathy
* Steroid myopathy
* Cervical spine injury, lesions, or large osteophytes
* Kerns-Sayers Syndrome
* Individuals unable to exercise independently
* Oculo-pharyngeal and other dystrophies
* Current use of anticholinergics:

bensodiazopin, antihistamines

* Myasthenia gravis
* Elimination of aspiration with posture during VFG
* Absent pharyngeal swallow on VFG
* Aspiration before or during the swallow (pre and intradeglutitive aspiration)
* Not completely tube feeding dependent

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204
Dates: Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reza Shaker, M.D., Principal Investigator — Professor and Chief, Division of Gastroenterology and Hepatology, Director, Digestive Disease Center, Medical College of Wisconsin; Jerilyn A. Logemann, Ph.D., Principal Investigator — Professor Department of Communication Sciences and Disorders, Ralph and Jean Sundin Professor of Communication Sciences and Disorders, Northwestern University
Locations (1):
- Medical College University of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Shaker R, Easterling C, Kern M, Nitschke T, Massey B, Daniels S, Grande B, Kazandjian M, Dikeman K. Rehabilitation of swallowing by exercise in tube-fed patients with pharyngeal dysphagia secondary to abnormal UES opening. Gastroenterology. 2002 May;122(5):1314-21. doi: 10.1053/gast.2002.32999. PMID 11984518
- See also: Division of Gastroenterology and Hepatology — http://www.mcw.edu